CLINICAL TRIAL: NCT07001306
Title: A Prospective Clinical Study of Long-term Effects of SCL-wearing on Corneal Neuromediators and Postoperative Rehabilitation After SMILE
Brief Title: Long-term Effects of SCL-wearing on Corneal Neuromediators and Postoperative Rehabilitation After SMILE
Acronym: SCL SMILE
Status: Completed | Type: Observational
Sponsor: yuhao shao (Other)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor-Investigator, yuhao shao, MD, Tongji University
Organization: Tongji University (Other)
Other Study IDs: SCL on SMILE visual quality; 202240131 (Other Grant/Funding Number: Shanghai Municipal Health Commission); YJXYS-B-009 (Other Grant/Funding Number: Shanghai Tenth People's Hospital); YNCR2C004 (Other Grant/Funding Number: Shanghai Tenth People's Hospital); 2023SQ03 (Other Grant/Funding Number: Shanghai Association of Chinese Integrative Medicine)
Record Dates: First submitted 2025-05-22; First posted 2025-06-03 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Contact Lens Complication; Small Incision Lenticule Extraction
Keywords: small incision lenticule extraction; neuromediators; visual quality; corneal nerve regeneration; soft contact lens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All samples were collected from participants with myopia who underwent SMILE surgery. The VisuMax femtosecond laser system (Carl Zeiss Meditec, Jena, Germany) was utilized with the following settings: a repetition rate of 500 kHz, pulse energy of 150 nJ, intended cap thickness of 110-120 μm, and optical zone of 6.0-6.8 mm. A circumferential incision width of 2 mm was made for lenticule dissection and extraction. The surgical procedures were performed by a single experienced surgeon (Dr. Zou). Following the SMILE surgeries, corneal stromal lenticules were transferred to Eppendorf tubes and stored at -80°C. for subsequent analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SCLs >10 years: myopia patients who wear SCL more than 10 years before Small Incision Lenticule Extraction
- SCLs ≤10 years: myopia patients who wear SCL for 10 years or less before Small Incision Lenticule Extraction
- NW: myopia patients who have not worn SCLs before Small Incision Lenticule Extraction

SUMMARY:
To investigate the effects of neuromediators in corneal stromal lenticules from patients with long-term soft contact lens (SCL) wear on corneal nerve regeneration and visual quality recovery following small incision lenticule extraction (SMILE).

DETAILED DESCRIPTION:
he prospective cohort study recruited 90 patients who underwent SMILE between June 2023 and June 2024. 90 eyes were categorized into three groups according to the duration of wearing SCL: the > 10 years group (25 eyes), the ≤ 10 years group (35 eyes), and the non-wear (NW) group (30 eyes). Pre- and post-operative assessments at 1, 3 and 6 months included corneal higher-order aberrations (HOAs), corneal optical density, tear film breakup time (BUT), corneal fluorescein staining, subepithelial corneal nerve fiber parameters, Ocular Surface Disease Index (OSDI), Quality of Vision (QOV) scores, and contrast sensitivity function (CSF). nerve growth factor (NGF), insulin-like growth factor binding protein-1 (IGFBP-1), mesencephalic astrocyte-derived neurotrophic factor (MANF), calcitonin gene-related peptide (CGRP) and substance P (SP) in stromal lenticules were quantified using ELISA. Multiple linear regression analysis was employed to evaluate the associations between SCL wear duration, mediator levels, and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years with stable refraction for at least two years;
* corrected distance visual acuity of 20/20 or better;
* no history of using rigid gas permeable lenses or orthokeratology (OK) lenses prior to examination

Exclusion Criteria:

- a history of moderate to severe dry eye as well as any ocular or systemic disease that would contraindicate laser refractive surgery.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with myopia who underwent SMILE surgery at Shanghai Tenth People's Hospital in Shanghai, China, from June 2023 to the present.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Quality of Vision (QOV) scores | baseline, 1 month, 3months, 6months
  It consists of 10 items related to visual symptoms, including glare, halo, radiating light, foggy vision, blurred vision, visual distortion, diplopia, visual fluctuation, difficulty in focusing and difficulty in depth perception. Each item consists of three dimensions: frequency, severity and degree of distress. Therefore, this questionnaire contains a total of 30 questions. The answers to the above three dimensions respectively include four options, namely frequency: never, occasionally, often, and frequently; Severity: None, mild, moderate, severe; Degree of distress: None, a little, some, very much. The corresponding scores for the four options are 0, 1, 2, and 3 respectively. The higher the score, the worse the visual quality
contrast sensitivity function | baseline, 1moth, 3 moths, 6 months
  Under sufficient correction conditions, dark adaptation lasted for 10 minutes. Using the CSV-1000 contrast sensitivity tester at a distance of 3 meters, under the conditions of bright vision (85 cd/m ²), bright glare (135 lx), dark vision (3 cd/m ²), and dark glare (28 lx) respectively, Test the highest CS level that can be distinguished at 3, 6, 12 and 18 c/d spatial frequencies one by one. At each spatial frequency, the examinee needs to point out the bar grid sight in the upper and lower two circular sight targets and report the direction of the bar grid. After the result is correct, gradually reduce the bar grid contrast until the examinee can no longer recognize it. The inverse of the lowest recognizable contrast at this time is the contrast sensitivity. Record in logarithmic units according to the grade value conversion table.
Corneal subepithelial nerve fibers | baseline, 1moth, 3 moths, 6 months
  In this study, the ACCMetrics V.2 software developed by the University of Manchester in the UK for the HRT confocal microscope of Heidelberg Company was used to conduct automatic quantitative analysis and data recording on three nerve fiber images at different positions selected in a single shoot. The parameters analyzed include corneal nerve fiber density (CNFD sterand/mm 2) and corneal nerve fiber length( CNFL, mm/mm 2), corneal nerve fiber area (CNFA mm2/mm 2), corneal nerve fiber width (CNFW mm ), etc. Each inspection is carried out by the same inspector to reduce subjective errors.
Corneal stromal lenticule Neuromediators | baseline
  Corneal neuromediators, including NGF(pg/mL), CGRP(pg/mL), SP(pg/mL), IGFBP-1(ng/mL), and MANF(pg/mL), which play pivotal roles in maintaining normal physiological functions of the cornea.
OSDI Questionnaire | baseline, 1moth, 3 moths, 6 months
  The impact of dry eye on the subjective symptoms of patients was evaluated from three dimensions: ocular symptoms, visual function, and environmental stimuli. There were a total of 12 items. Each symptom was divided into 5 levels according to the degree and occurrence frequency: 0 was considered as none. 1 point occurs sometimes; 2 minutes occurs approximately half of the time; 3 points occur frequently; 4 points occur continuously. The final OSDI score = the total of all scores ×100/ (the total number of assessment questions ×4), with a total score ranging from 0 to 100.

SECONDARY OUTCOMES:
Tear film stability | baseline, 1moth, 3 moths, 6 months
  Including corneal fluorescein staining score and tear film break-up time examination.
  Corneal fluorescein staining score The corneal fluorescein staining was observed in different regions under a cobalt blue filter and scored. The cornea was divided into three regions: upper, middle and lower. Scores were given based on the fluorescein staining of the corneal epithelium in each region. No staining was scored as 0 points, 1 point for 1 to 30 staining points, 2 points for more than 30 staining points and no fusion of the staining points, and 3 points for the presence of corneal patellar staining fusion, filamentous substances and ulcers, etc. The total score is 9 points.
  Tear film break-up time Instruct the patients to look straight ahead, observe with a slit lamp and cobalt blue filter, and measure the time when dry spots first appear on the cornea after one involuntary blinking movement with a stopwatch. Each patient is measured three times, and the average of the three measurements i
Corneal Aberration | baseline, 1moth, 3 moths, 6 months
  Preoperative corneal aberration measurements were performed using a Scheimpflug tomography system (Pentacam; Oculus GmbH, Wetzlar, Germany). Images of the highest quality (designated as OK) were selected for analysis. The coefficients for a standardized diameter of 8 ?mm were examined, followed by an assessment of the clinical significance of total higher-order aberrations (HOA, mm), spherical aberration (Z4, 0, mm), horizontal coma (Z3, 1, mm), vertical coma (Z3, -1, mm), horizontal trefoil (Z3, 3, mm), and oblique trefoil (Z3, -3, mm) in relation to visual quality.
Corneal Densitometry | baseline, 1moth, 3 moths, 6 months
  The Pentacam HR was used to collect data on corneal densitometry values, which were expressed in grayscale units (GSUs), playing a crucial role in quantifying corneal clarity by monitoring transient haze-like reactions. The cornea was divided into four annular zones (0-2 mm, 2-6 mm, 6-10 mm, and 10-12 mm), each exhibiting distinct corneal densitometry values. Based on the anatomical layers of the cornea at different depths, it consists of four layers: a superficial anterior layer of 120 μm, a posterior layer located within the innermost part of the cornea measuring 60 μm; central layers calculated by subtracting thickness of the anterior and posterior layers from the total layer thickness; and a total layer. Corneal densitometry values were measured in the 0-2 mm and 2-6 mm to correspond to the corneal optical zone diameter of SMILE.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No